CLINICAL TRIAL: NCT02892747
Title: Impact of Dietetics Education Focused on Prevention of Malnutrition, on Reducing Morbidity and Improving Life Quality of Patients With Chronic Heart Failure (CHF): A Randomized Controlled Multicenter Clinical Trial
Brief Title: Dietetics Education Focused on Malnutrition Prevention
Acronym: NUTRICOEUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K140703
Record Dates: First submitted 2016-07-31; First posted 2016-09-08 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Chronic Heart Failure (CHF)
Keywords: Chronic Heart Failure (CHF); Dietetics education; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Program for prevention of malnutrition (Experimental): In addition to the usual nutritional assessment, the patients in the experimental arm benefit of a personalized educational program for prevention of malnutrition. This program aims to monitor energy and protein intake in addition to managing sodium intake, notably by offering personalized menu ideas and recipes.
  Interventions: Behavioral: Educational Program
- Control (No Intervention): In the control arm, patients are followed-up by the cardiologist and the nutritionist, and did not benefit of the personalized educational program for prevention of malnutrition.

INTERVENTIONS:
Behavioral: Educational Program
  Arms: Educational Program for prevention of malnutrition

SUMMARY:
The intervention tested in this research project aims to reduce the unplanned hospitalizations in CHF patients by preventing the malnutrition using a personalized dietetic education program. This new program provides concrete solutions to patients by offering balanced menu ideas, adapted to their tastes and social-cultural habits, and a panel of recipes easy to make, inexpensive and tasty (despite the lack of salt). This new educational program should improve the dietary behavior of patients and reinforce the importance of dietary guidance in support of the CHF.

DETAILED DESCRIPTION:
Context: The Chronic Heart Failure (CHF) is a major public health problem in terms of frequency, mortality and costs. The care integrates a low-salt diet to reduce fluid retention and cardiac decompensation. A large observational study (ODIN) shows the effectiveness of the Patient's Therapeutic Education program (PTE which provides learning management sodium intake by the intervention of a dietician, I-CARE) on reducing mortality. But prognosis of CHF remains serious leading to many hospitalizations. The nutritional status of patients with CHF is threatened by inadequate energy intake in connection with the low sodium diet and the rest energetic cost (REC). Malnutrition increases the risk of hospitalization because it causes an immune deficiency responsible for infections, bones weakness and impaired cognitive function.

Hypotheses: The investigators postulate that an educational diet focusing on prevention of malnutrition would reduce morbidity and improve quality of life for patients with CHF. For this, the investigators propose a new educational method: adding a personalized program monitoring energy and protein intake in addition to managing sodium intake, notably by offering personalized menu ideas and recipes.

Main objective: Demonstrate that a dietetic education program involving the prevention of malnutrition and managing sodium intake is more effective than the usual dietetic education (based only on management of sodium intake) on the frequency of unplanned hospitalizations (all causes ) at 6 months in CHF patients.

Secondary Objectives: Demonstrate the superiority of the dietetic education program involving the prevention of malnutrition and managing sodium intake over the usual dietetic education, by improving the nutritional status, the quality of life, the survival, the adherence to dietary recommendations and the reduction of hospitalizations for cardiac decompensation, the burden associated with low sodium diet and the costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years old and over.
* Patients with Chronic Heart Failure regardless of its severity stage: stage I to IV according to the New York Heart Association Classification (NYHC), and its age.
* Patients having at least a cardiac failure on the last two years.
* BMI ≥ 18,5 (≥ 21 if Age ≥ 70 years).
* Patients with a prescription of dietary salt restriction, regardless of the amount of salt recommended.
* Patients benefiting from the Patient Therapeutic Education Program (ICARE) focusing on managing sodium intake.
* Patients informed of the study, and have given their oral non opposition.
* Patients insured by a social security.

Exclusion Criteria:

* Severe comorbidity (outside the CHF) affecting the prognosis at 3 months
* Living in nursing homes or in housing home where it is difficult to manage their feed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Estimated)
Dates: Start 2016-09; Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
The number, duration, reason of hospitalization will be reported in a tracking booklet that will be given to the patient the day of his/her inclusion | 6 months after randomization

SECONDARY OUTCOMES:
Sodium intake will be evaluated by dietary survey on 24-hour recall and also by a rich-salt food frequency questionnaire | 8th day, 1 month, 2 months, 3 months, 4 months, 5 months and 6 months
Protein supply (g / day) will be assessed by dietary survey on 24-hour recall and also by a food frequency questionnaire. | 8th day, 1 month, 2 months, 3 months, 4 months, 5 months and 6 months
Energy intake (Kcal/day)will be assessed by dietary survey on 24-hour recall and also by a food frequency questionnaire. | 8th day, 1 month, 2 months, 3 months, 4 months, 5 months and 6 months
EuroQol five dimensions questionnaire (EQ-5D) | 6 months after randomization
Minnesota Living With Heart Failure Questionnaire (MLHFQ) | 6 months after randomization
Questionnaire "burden of diet" | 6 months after randomization
The compliance of dietary recommendations will be assessed by a tracking booklet in which food dietary recommendations will be reported | 8th day, 1 month, 2 months, 3 months, 4 months, 5 months and 6 months
The unplanned hospitalizations frequency for cardiac decompensation | 6 months after randomization
Death (cardiac cause included) | 8th day, 1 month, 2 months, 3 months, 4 months, 5 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Véronique BENEDYGA, Nutritionist, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Nicol SM, Carroll DL, Homeyer CM, Zamagni CM. The identification of malnutrition in heart failure patients. Eur J Cardiovasc Nurs. 2002 Jun;1(2):139-47. doi: 10.1016/s1474-5151(02)00005-1. PMID 14622767
- [Background] Arcand J, Floras V, Ahmed M, Al-Hesayen A, Ivanov J, Allard JP, Newton GE. Nutritional inadequacies in patients with stable heart failure. J Am Diet Assoc. 2009 Nov;109(11):1909-13. doi: 10.1016/j.jada.2009.08.011. PMID 19857633
- [Background] Curtis JP, Selter JG, Wang Y, Rathore SS, Jovin IS, Jadbabaie F, Kosiborod M, Portnay EL, Sokol SI, Bader F, Krumholz HM. The obesity paradox: body mass index and outcomes in patients with heart failure. Arch Intern Med. 2005 Jan 10;165(1):55-61. doi: 10.1001/archinte.165.1.55. PMID 15642875
- [Background] Beck CA, Shah S. Research on health-related quality of life and cardiac conditions. Home Healthc Nurse. 2012 Jan;30(1):54-60. doi: 10.1097/NHH.0b013e31823aa740. PMID 22173621
- [Background] Ferrante D, Varini S, Macchia A, Soifer S, Badra R, Nul D, Grancelli H, Doval H; GESICA Investigators. Long-term results after a telephone intervention in chronic heart failure: DIAL (Randomized Trial of Phone Intervention in Chronic Heart Failure) follow-up. J Am Coll Cardiol. 2010 Jul 27;56(5):372-8. doi: 10.1016/j.jacc.2010.03.049. PMID 20650358